CLINICAL TRIAL: NCT05277818
Title: Clinical Follow-up of the DIVA® Device in Lumbar Disc Herniation Surgery
Brief Title: Post-marketing Clinical Follow-up of the Medical Device DIVA®
Status: Recruiting | Type: Observational
Sponsor: SC Medica (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A02667-34
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with medical device DIVA®: Adult patient, operated for at least 12 months, having had surgery for a degenerative or traumatic mono-segmental lumbar disc herniation, without any other associated pathology, operated with DIVA® implant
  Interventions: Procedure: Surgery lumbar disc herniation
- Patient without medical device DIVA®: Adult patient, operated for at least 12 months, having had surgery for a degenerative or traumatic mono-segmental lumbar disc herniation, without any other associated pathology, operated without DIVA® implant
  Interventions: Procedure: Surgery lumbar disc herniation

INTERVENTIONS:
Procedure: Surgery lumbar disc herniation — Surgery for a degenerative or traumatic mono-segmental lumbar disc herniation

SUMMARY:
Observational, ambispective, longitudinal, comparative, open, multicentric study.

The main objective is to compare the performance of care in patients operated with and without DIVA®.

DETAILED DESCRIPTION:
The primary endpoint is the reoperation for any cause (excluding trauma) on the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, having undergone surgery for a degenerative or traumatic mono-segmental lumbar disc herniation, without any other associated pathology, operated with or without a DIVA® implant;
* Patient operated for at least 12 months;
* Patient able to understand the information related to the study;
* Patient having indicated his/her non-opposition to the collection of his/her personal data.

Exclusion Criteria:

* History of pathologies, malformations or surgical interventions on the spine;
* Patient belonging to the first 30 operated by the surgeon with the DIVA® implant;
* Protected patient (under legal protection, or deprived of liberty by judicial or administrative decision);
* Patient not benefiting from a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with the DIVA® device operated in the study centers for at least 12 months (with the exception of the first 30 operated by practitioner, to take into account the learning curve), as well as all patients operated on over a period similar before the installation of DIVA® in the establishment, will receive the information note of the study. if the patient agrees to participate to the study, patient's data will be collected on a case report form.
Sampling Method: Probability Sample
Enrollment: 822 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Rates of patients requiring reoperation for any cause (excluding trauma) on the lumbar spine 5 years postoperatively. | 5 years
  The main analysis will compare the rates of patients requiring reoperation due to any cause (excluding trauma) on the lumbar spine 5 years after surgery between the group with DIVA® and the group without DIVA®, using a Chi-square test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Civils de Colmar, Colmar, France

IPD SHARING:
Plan to Share IPD: No